CLINICAL TRIAL: NCT06954402
Title: A Novel Human Laboratory Model of Resilience Among Individuals With Opioid Use Disorder
Brief Title: Resilience Among Individuals With Opioid Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00438915; K08DA058057 (NIH)
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
Keywords: opioids; opioid use disorder; stress
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress-First Sequence (Experimental): Participants in this arm will first undergo the stress condition using the Maastricht Acute Stress Test (MAST) and then complete the non-stress condition (NST) in a subsequent session.
  Interventions: Behavioral: Acute Stress Intervention (MAST-based); Behavioral: Non-Stress Intervention (NST-based)
- Non-Stress-First Sequence (Experimental): Participants in this arm will first complete the non-stress condition (NST) and then undergo the stress condition using the Maastricht Acute Stress Test (MAST) in a subsequent session.
  Interventions: Behavioral: Acute Stress Intervention (MAST-based); Behavioral: Non-Stress Intervention (NST-based)

INTERVENTIONS:
Behavioral: Acute Stress Intervention (MAST-based) — This intervention uses the Maastricht Acute Stress Test (MAST) to induce an acute stress response. Participants are exposed to standardized stress tasks while performing laboratory-based assessments of cognitive, emotional, and control aspects of resilience.
Behavioral: Non-Stress Intervention (NST-based) — In this control intervention, participants complete the same battery of laboratory tasks without exposure to the acute stressor.

SUMMARY:
The goal of this clinical trial is to develop a human laboratory model of resilience in people with opioid use disorder (OUD). The investigators aim to learn if objective tasks that measure cognitive, emotional, and control aspects of resilience match up with self-reported resilience during stress and non-stress situations.

DETAILED DESCRIPTION:
This study is an outpatient, within-subject, randomized controlled trial designed to develop and validate a novel laboratory-based model for assessing resilience in individuals with opioid use disorder (OUD). The study employs a dual-condition design where participants complete two experimental sessions administered in a randomized order: one under a stress condition and under a non-stress condition. In each session, participants will perform a series of standardized laboratory tasks aimed at evaluating cognitive, emotional, and control aspects of resilience. Objective measures (e.g., task performance data and physiological indices) and subjective ratings of stress reactivity will be collected to capture both behavioral and self-perceived responses.

ELIGIBILITY:
Inclusion Criteria:

1. Can provide informed consent and can comply with study procedures
2. Adults aged ≥18 years
3. Meet Diagnostic and Statistical Manual (DSM-5) criteria for current opioid use disorder or are currently receiving pharmacotherapy for the treatment of OUD (e.g. methadone or buprenorphine maintenance treatment [remission])
4. Urine sample that tests positive for opioids
5. Test negative for pregnancy at screening (females only)

Exclusion Criteria:

1. Being pregnant or breastfeeding
2. Significant mental health or physical disorder, or life circumstances, that is judged by the investigators to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Trait Resilience as assessed by Connor-Davidson Resilience Scale 25 (CD-RISC-25) | Immediately after completing the task
  Instrument: Connor-Davidson Resilience Scale 25 Score Range: 0-100 Interpretation: Higher scores indicate greater resilience.
Cognitive Flexibility: Stroop Color-Word Test reaction time | Immediately after completing the task
  Instrument: Stroop Color-Word Test Unit: Milliseconds (ms) Interpretation: Higher values = slower performance (worse)
Emotional Flexibility: Emotional Stroop Task reaction time | Immediately after completing the task
  Instrument: Emotional Stroop Task Unit: Milliseconds (ms) Interpretation: Higher values = slower performance (worse).
Perceived Controllability (Controllable) assessed by Social Controllability Task (SCT) | Immediately after completing the task
  Instrument: Social Controllability Task Description: Participants ratings on a 0-100% sliding scale. Interpretation: Higher scores indicate greater perceived control.

SECONDARY OUTCOMES:
Subjective Effects of Stress as assessed by the Subjective Effects Visual Analog Scale (VAS) Battery | Immediately after completing the task
  Instrument: Subjective Effects Visual Analog Scale (VAS) Battery Instrument: VAS (0-100 mm) Interpretation: Higher scores indicate greater intensity of each subjective state.
Heart Rate | Immediately after completing the task
  Unit: Beats per minute (bpm) Interpretation: Higher = increased arousal
Systolic Blood Pressure | Immediately after completing the task
  Unit: mmHg Interpretation: Higher = greater pressure.
Diastolic Blood Pressure | Immediately after completing the task
  Unit: mmHg Interpretation: Higher = greater pressure.
Opioid Demand Breakpoint as assessed by the Hypothetical Purchase Task | Immediately after completing the task
  Instrument: Hypothetical Purchase Task Range: $0-$500 Interpretation: Higher = greater demand.

CONTACTS AND LOCATIONS:
Overall Officials: Suky Martinez, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Bayview Medical Campus, Baltimore, Maryland, United States